CLINICAL TRIAL: NCT07288073
Title: A Feasibility Study of Tumor Infiltrating Lymphocytes in Cutaneous Squamous Cell Carcinoma and Merkel Cell Carcinoma
Brief Title: TIL Therapy in cSCC and MCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karam Khaddour (Other)
Collaborators: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Karam Khaddour, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-394
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Merkel Cell Carcinoma; Metastatic Cutaneous Squamous Cell Carcinoma; Skin Cancer
Keywords: Cutaneous Squamous Cell Carcinoma; Merkel Cell Carcinoma; Metastatic Cutaneous Squamous Cell Carcinoma; Skin Cancer
MeSH Terms: conditions — Carcinoma, Merkel Cell; Skin Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: CSCC Autologous TIL Therapy (Experimental): 10 participants with CSCC will complete:
  * Screening visit
  * Surgical procedure to collect tissue, called TIL harvest
  * Baseline visit
  * Days -5 through -1: Predetermined dose of Lymphodepleting Chemotherapy, Fludarabine, 1x daily
  * Days -5 and -4: Predetermined dose of Lymphodepleting Chemotherapy, Cyclophosphamide, 1x daily
  * Day 0: TIL infusion
  * Days 0, 1, 2, 3, 4, and 14: Predetermined dose of IL-2 1x daily for up to 6 doses
  * Imaging at weeks 6 and 12
  * End of treatment visit with imaging
  * Long term follow up every 3 months for up to 3 years
  Interventions: Biological: LN-145; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Interleukin-2
- Cohort B: MCC Autologous TIL Therapy (Experimental): 4 participants with MCC will complete:
  * Screening visit
  * Surgical procedure to collect tissue, called TIL harvest
  * Baseline visit
  * Days -5 through -1: Predetermined dose of Lymphodepleting Chemotherapy, Fludarabine, 1x daily
  * Days -5 and -4: Predetermined dose of Lymphodepleting Chemotherapy, Cyclophosphamide, 1x daily
  * Day 0: TILs infusion
  * Days 0, 1, 2, 3, 4, and 14: Predetermined dose of IL-2 1x daily for up to 6 doses
  * Imaging at weeks 6 and 12
  * End of treatment visit with imaging
  * Long term follow up every 3 months for up to 3 years
  Interventions: Biological: LN-145; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Interleukin-2

INTERVENTIONS:
Biological: LN-145 — Autologous tumor-infiltrating lymphocytes via intravenous (into the vein) infusion per protocol
  Other Names: Autologous Tumor Infiltrating Lymphocytes
Drug: Cyclophosphamide — Antineoplastic drug, multi-dose vial, per institutional standards
  Other Names: Cytoxan; Cyclophosphamide-OE
Drug: Fludarabine — Nucleotide metabolic inhibitor, single-use vial, via intravenous infusion per institutional standards
  Other Names: Fludarabine Phosphate
Biological: Interleukin-2 — Recombinant, human glycoprotein, single-use vial, via intravenous infusion per protocol
  Other Names: Aldesleukin; Proleukin; IL-2

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of a tumor-infiltrating lymphocyte (TIL) cellular therapy, also called LN-145 or lifileucel, and chemotherapy in combination with Interleukin-2 (IL-2) to find out what effects, if any, the combination has on participants with Cutaneous squamous cell carcinoma (CSCC) or Merkel Cell Carcinoma (MCC) who were previously treated with immunotherapy.

The names of the study interventions involved in this study are:

* Tumor Infiltrating Lymphocytes (a type of cellular therapy)
* Fludarabine and Cyclophosphamide (types of standard of care chemotherapy drugs)
* Interleukin-2 (a type of recombinant, human glycoprotein)

DETAILED DESCRIPTION:
This is an open-label, multi-cohort, non-randomized, single-center, phase 2 clinical trial testing the safety and effectiveness of a tumor-infiltrating lymphocyte (TIL) cellular therapy, also called LN-145 or lifileucel, and chemotherapy in combination with Interleukin-2 (IL-2) to find out what effects, if any, the combination has on participants with Cutaneous squamous cell carcinoma (CSCC) or Merkel Cell Carcinoma (MCC) who were previously treated with immunotherapy.

Lymphocytes are a part of the immune system that help fight infection and prevent and fight cancers. TIL cells are grown in a specialized laboratory with the goal of making more of them so that the TIL cells better recognize and kill cancer cells when administered again into the body.

The U.S. Food and Drug Administration (FDA) has approved Fludarabine and Cyclophosphamide as standard-of-care lymphodepleting chemotherapy medications.

The U.S. FDA has not approved TIL therapy, Lifileucel plus IL-2, for CSCC or MCC, but it has been approved for the treatment of another type of skin cancer, advanced melanoma.

The research study procedures include screening for eligibility, in-clinic visits, blood tests, urine tests, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, or Positron Emission (PET) scans, X-rays, electrocardiograms (ECGs), echocardiograms (ECHOs), Cardiac stress test, lung function test, bone marrow biopsies and aspirations.

It is expected that about 14 people will take part in this research study.

Iovance Biotherapeutics, Inc. is supporting this research study by providing the study therapy, IL-2 and funding.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent, which includes understanding that there may be a need for intensive supportive care measures during the study and assessing willingness to undergo such measures, and written authorization for use and disclosure of protected health information.
* Patients must be ≥ than 18 years of age at the time of signing the informed consent form.
* Patients must have histologically or pathologically confirmed diagnosis of CSCC or MCC. Note: Mixed histology is allowed. Note: Neuroendocrine cancer that is clinically considered to be related to a cutaneous primary (MCC) or induced by sun damage (per investigator assessment) is allowed.
* Patients must have unresectable, recurrent, or metastatic disease.
* Patients must have a documented radiographic or clinical disease progression after treatment with ICI (including anti-PD-1 and anti-PD-L1) if it is used in the palliative setting. In patients who received ICI in the neoadjuvant or adjuvant setting, recurrence should have occurred within 6 months from the last treatment with ICI.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 in the investigator's opinion (Appendix B).
* Patients must have at least 1 resectable lesion (or aggregate lesions) with an expected minimum of 1.5 cm diameter in the short axis for TIL production. Note: If a lesion that is considered for TIL harvest is within a previously irradiated field, the lesion must have demonstrated radiographic or clinical progression prior to harvest, and the irradiation must have been completed at least 6 months prior to enrollment.
* Patients must be expected to have at least 1 remaining measurable lesion as defined by RECIST v1.1 or evaluable (radiographically or on clinical examination) following tumor harvest for TIL manufacturing and production that is documented at screening with the following considerations:

  * Lesions in a previously irradiated areas should not be selected as target lesions unless progression has been demonstrated in those lesions and the irradiation has been completed at least 6 months prior to enrollment.
  * Patients who have only one site of disease may be enrolled if they have a lesion th can be partially resected for TIL harvest, and the remaining portion of the lesion is measurable or evaluable.
* Patients must have the following hematologic parameters:

  * Absolute neutrophil count (ANC) ≥ 1000/mm3
  * Hemoglobin ≥ 8.0 g/dL and have not received transfusion of packed red blood cells within 7 days.
  * Platelet count ≥ 100,000/mm3
* Patients must have an adequate organ function with the following laboratory test values:

  * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal (ULN); and for patients with liver metastases ≤ to 5 times ULN.
  * Total bilirubin ≤ 2 mg/dL; patients with Gilbert's Syndrome ≤ to 3 mg/dL.
  * Estimated creatinine clearance (eCrCl) ≥ 40 mL/min using the Cockcroft-Gault formula at Screening.
* Patients must have a left ventricular ejection fraction (LVEF) ≥ 45% and be New York Heart Association (NYHA) Class 1 or 2. A cardiac stress test is required for patients who have significant ischemic heart disease, or clinically significant unstable arrythmias; the cardiac stress test must demonstrate no irreversible wall movement abnormality. Patients with an abnormal cardiac stress test may be enrolled if they have adequate ejection fraction and cardiology clearance.
* Patients must have adequate pulmonary function within 2 months from enrollment.

Patients require pulmonary function testing (PFT) if they have any of the following:

* History of cigarette smoking of ≥ 20 pack-years
* Ceased smoking within the past 2 years or still smoking.
* History of chronic obstructive pulmonary disease (COPD)
* Any signs or symptoms of significant respiratory dysfunction.

Post-bronchodilator required pulmonary test results:

* Forced expiratory volume (FEV1)/ forced vital capacity (FVC) > 70%. Or
* FEV1 > 50% of predicted normal value. Note: If a patient is unable to perform reliable spirometry due to abnormal upper airway anatomy (i.e., tracheostomy), a 6-minute walk test may be used to assess pulmonary function. Patients must be able to walk a distance at least 80% of predicted for age and sex with no evidence of hypoxia at any point during the test (i.e., saturation of peripheral oxygen [SpO2] must remain ≥ 89%).

  * Patients must have completed or discontinued systemic therapy ≥ 21 days prior to tumor harvest. Note: Patients are allowed to have palliative radiation or systemic therapy after tumor harvest and before NMA-LD but there should be at least 7 days between discontinuation of palliative treatment and start of NMA-LD.
  * Patients must have recovered from all prior anticancer TRAEs to Grade ≤ 1 (per CTCAE v5.0) with the exceptions of vitiligo, alopecia or neuropathy. Patients with irreversible toxicity that are properly managed (such as with endocrinopathy treatment with hormone replacement therapy) may qualify for the study regardless of grade of TRAEs.
  * Patients of childbearing potential or those with partners of childbearing potential must be willing to practice an approved method of highly effective birth control during treatment and for 12 months after receiving all protocol-related therapy (Appendix C). Additionally, males may not donate sperm and females may not donate eggs during the required contraception period.

Approved methods of birth control include:

* Combined (estrogen- and progesterone- containing) hormonal birth control associated with inhibition of ovulation: oral, intravaginal, transdermal.
* Progesterone-only hormonal birth control associated with inhibition of ovulation:

oral, injectable, implantable.

* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomy
* True absolute sexual abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar ovulation, symptothermal, post-ovulation methods) is not acceptable.

Exclusion Criteria:

* Have a history of allogenic organ transplant.
* Have symptomatic untreated brain metastases. Patients with brain metastases may be enrolled with the following considerations:

  * Patients with asymptomatic brain metastases that are treated and have been stable for at least 7 days may be enrolled.
  * Patients with historically or recently treated brain metastases will be considered for enrollment if the patient is clinically stable for ≥ 2 weeks, and the patient does not require ongoing corticosteroid treatment (>10 mg/day prednisone or its equivalent).
  * Patients who undergo tumor harvest prior to disease progression and develop symptomatic brain metastases after tumor harvest should have receive appropriate treatment for ≥ 2 weeks and not require corticosteroids (>10 mg/day or its equivalent) at the start of NMA-LD (Day -5).
* Require systemic steroid therapy >10 mg/day prednisone or its equivalent. Patient receiving steroids as replacement therapy for adrenocortical insufficiency are not excluded.
* Have evidence of any active viral, bacterial, or fungal infection requiring ongoing systemic treatment.
* Are pregnant or breastfeeding. Female patients of childbearing potential must have a negative beta human chorionic gonadotropin (B-HCG) test at Screening (Appendix C).
* Have active medical illness that in the opinion of the investigator would pose increased risk for study participation, such as systemic infections, coagulation disorders, or other active major medical illnesses of the cardiovascular, respiratory, or immune system.
* Have received a live or attenuated vaccination within 28 days prior to the start of NMALD.
* Have any form of primary immunodeficiency (e.g., severe combined immunodeficiency disease [SCID] or acquired immune deficiency syndrome [AIDS]).
* Have a history of allogenic stem cell transplant, or active hematological malignancy (such as chronic lymphocytic leukemia or lymphoma).
* Have a history of hypersensitivity to any component of the study drugs. TIL should not be administered to patients with a known hypersensitivity to any component of the autologous TIL product formulation including, but not limited to, any of the following:

  * NMA-LD (cyclophosphamide, mesna, and fludarabine)
  * Proleukin, aldesleukin, IL-2
  * Antibiotics of the aminoglycoside group. These patients may be eligible if current hypersensitivity has been excluded.
  * Any component of the TIL product formulation, including dimethyl sulfoxide (DMSO), human serum albumin (HSA), IL-2, or dextran-40
* Have had another primary malignancy within the previous 1 year (except for malignancies that do not require treatment or have been curatively treated, and do not pose a significant risk of recurrence including, but not limited to in situ carcinoma of the cervix, early stage skin cancer, including non-melanoma skin cancer; ductal carcinoma in situ (DCIS) or lobular carcinoma in the situ (LCIS) of the breast; intraductal carcinoma of the breast that has been treated with curative intent including patients who are on adjuvant hormonal treatment, prostate cancer with Gleason score ≤ to 6; or superficial bladder cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-09-29 (Estimated); Study Completion 2029-06-29 (Estimated)

PRIMARY OUTCOMES:
Tumor-infiltrating lymphocyte (TIL) Production | TIL infusion will be performed at day 0 of the study.
  Tumor-infiltrating lymphocyte (TIL) production is defined by the successful tumor harvest that leads to a manufacturing of a TIL product that contains ≥ 1 x 10^9 cells.
Tumor-infiltrating lymphocyte (TIL) Administration | Evaluated up to 24 hours from TIL infusion (day 0) as IL-2 first dose will be administered with in 12-24 hours from TIL infusion.
  TIL administration is defined by the administration of NMA-LD, complete infusion of TIL therapy and at least 1 dose of interleukin-2 (IL-2).
Incidence of Grade ≥3 treatment-emergent adverse events (TEAEs) | Adverse events will be collected until 30 days post treatments. The study does not have a fixed treatment duration as defined in the protocol section 5.5.
  TEAEs will determined on the Common Toxicity Criteria for Adverse Events Version 5.0 (CTCAEv5) as reported on case report forms.

SECONDARY OUTCOMES:
objective response rate (ORR) | Participants will be followed throughout the course of the trials for 3 years from the time of the end of treatment visit. The study does not have a fixed treatment duration as defined in the protocol section 5.5.
  ORR is defined as the proportion of participants receiving TIL therapy who achieve a best response of either complete response (CR) or partial response (PR) based on RECIST 1.1. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
progression-free survival (PFS) | Participants will be followed for 3 years from the end-of-treatment visit. The study does not have a fixed treatment duration, as specified in Section 5.5 of the protocol.
  PFS based on Kaplan-Meier method is defined as the time from study enrollment to the earlier of disease progression (RECIST 1.1) or death. The follow-up of participants who neither progress nor die will be censored at the date of the last follow-up. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
duration of response (DoR) | Participants will be followed for 3 years from the end-of-treatment visit. The study does not have a fixed treatment duration, as specified in Section 5.5 of the protocol.
  DOR is defined as the time from the first documentation of an objective response, either complete response (CR) or partial response (PR), to the time of disease progression or death, whichever occurs first. The follow-up of participants who have neither progressed nor died will be censored at the date of last follow-up. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
overall survival (OS) | Participants will be followed for 3 years from the end-of-treatment visit. The study does not have a fixed treatment duration, as specified in Section 5.5 of the protocol.
  Overall survival (OS) based on the Kaplan-Meier method is defined as the time from randomization to death. Participants alive are censored at the last date of contact (including lost-to-follow-up) or at the date of withdrawal of consent, if relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Karam Khaddour, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu